CLINICAL TRIAL: NCT05229198
Title: ALBATROSS Study: International Multicenter Study for Prospective Validation of Imaging Biomarkers Calculated at Vascular Habitats of High-grade Gliomas
Acronym: ALBATROSS
Status: Completed | Type: Observational
Sponsor: Juan M Garcia-Gomez (Other)
Collaborators: Oslo University Hospital (Other); Azienda Ospedaliero-Universitaria di Parma (Other); Hospital Clinic of Barcelona (Other); Hospital Vall d'Hebron (Other); Hospital de la Ribera (Other); Hospital de Manises (Other); Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Sponsor-Investigator, Juan M Garcia-Gomez, Main Researcher. Head of Biomedical Data Science Lab at UPV, Universitat Politècnica de València
Organization: Universitat Politècnica de València (Other)
Other Study IDs: ALBATROSS Study
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2022-02

CONDITIONS: Astrocytoma, Grade IV
Keywords: Astrocytoma, Grade IV; Glioblastoma; Glioblastoma IDH wildtype; Astrocytoma IDH mutant; Glioblastoma IDH mutant; High-grade glioma
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This Clinical study is framed in the ALBATROSS Project: Clinically validated decision support system based on pixel level Artificial Intelligent models for deciding treatment in glioblastoma.

The prospective multicenter international dataset compiled during the ALBATROSS project will include a cohort up to 300 new patients diagnosed with GB after June 1, 2020. Longitudinal images (T1, T2, T1c, FLAIR, PWI-DSC and DWI at least), complete molecular profiling, primary and secondary lines of treatment and clinical conditions will be included for each patient.

DETAILED DESCRIPTION:
The Hypothesis under study in this project is:

Therapeutic decision making during clinical management of patients with glioblastoma may benefit from delineating functional habitats at pixel level relative to growth, proliferation, infiltration and angiogenesis

The Overall Scientific Objectives of the research proposal are to:

OSO1. Delineate functional habitats from multiparametric MRI relative to the growth, proliferation, infiltration and angiogenesis at the enhanced tumor and infiltrated peripheral edema OSO2. Demonstrate that functional habitats at enhanced tumors and infiltrated peripheral edema show structural, cellular and molecular differences related to the heterogeneity of the tumor region and are compatible with mathematical models of glioma growth and infiltration OSO3. Determine the in-vivo molecular sub-type of patients with glioblastoma from image biomarkers in functional habitats OSO4. Identify groups of patients with glioblastoma presenting positive therapeutic response in terms of longer survival using image biomarkers from functional habitats OSO5. Position ONCOhabitats as a clinical decision support system for the management of patients with glioblastoma

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with astrocytoma grade IV WHO with histopathological/genetic confirmation who undergo the Stupp treatment
* Age > 18 years at diagnosis
* Patients with access to complete preoperative, postoperative and follow up MRI studies, including:

  * Pre gadolinium T1-weighted MRI
  * Post gadolinium T1-wighted MRI
  * T2-weighted MRI
  * Fluid-Attenuated Inversion Recovery (FLAIR)
  * Dynamic Susceptibility Contrast (DSC) T2*-weighted perfusion sequences
  * Diffusion Weighted Imaging (DWI)
* Patients who undergo surgery with the possibility to collect samples from different regions of the tumor

Exclusion Criteria:

* Patient with congestive heart failure within 6 months prior to study entry (New York Heart Association >= Grade 3)
* Uncontrolled or significant cardiovascular disease, including:

  * Myocardial infarction and transient ischemic attack or stroke within 6 months prior to enrollment
  * Uncontrolled angina within 6 months
  * Diagnosed or suspected congenital long QT syndrome
  * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
  * Clinically significant abnormality on electrocardiogram (ECG)
* Pulmonary disease including or greater than grade 2 dyspnea or laryngeal edema, grade 3 pulmonary edema or pulmonary hypertension according to CTCAE 4.03

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients diagnosed with astrocytoma grade IV WHO with histopathological/genetic confirmation who undergo the Stupp treatment
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of inclusion (date of first MRI) until the date of death, assessed up to 48 months
  Overall Survival is defined as the time from the first presurgical MRI is taken to the patient (MR0) to death

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From date of inclusion (date of first MRI) until the date of documented tumor progression, assessed up to 48 months
  Progression Free Survival is defined as the time from the first presurgical MRI is taken to the patient to the detection of tumor relapse

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Politècnica de València, Valencia, Valencia, Spain